CLINICAL TRIAL: NCT02858401
Title: A Phase 1b, Randomized, Blinded, Placebo-Controlled Dose-Escalation Study of the Safety and Biological Activity of GS-9620 in HIV-1 Infected, Virologically Suppressed Adults
Brief Title: Safety and Biological Activity of Vesatolimod in HIV-1 Infected, Virologically Suppressed Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-382-1450
Record Dates: First submitted 2016-07-26; First posted 2016-08-08 (Estimated); Results first posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — vesatolimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Vesatolimod 1 mg (Cohort 1) (Experimental): Vesatolimod 1 mg for 71 days, while continuing their existing ARV regimen
  Interventions: Drug: Vesatolimod; Drug: ARV regimen
- Vesatolimod 2 mg (Cohort 2) (Experimental): Vesatolimod 2 mg for 71 days, while continuing their existing ARV regimen
  Interventions: Drug: Vesatolimod; Drug: ARV regimen
- Vesatolimod 4 mg (Cohort 3) (Experimental): Vesatolimod 4 mg for 71 days, while continuing their existing ARV regimen
  Interventions: Drug: Vesatolimod; Drug: ARV regimen
- Vesatolimod 6 mg (Cohort 4) (Experimental): Vesatolimod 6 mg for 127 days, while continuing their existing ARV regimen
  Interventions: Drug: Vesatolimod; Drug: ARV regimen
- Vesatolimod 8 mg (Cohort 5) (Experimental): Vesatolimod 8 mg for 127 days administered following overnight fasting, while continuing their existing ARV regimen
  Interventions: Drug: Vesatolimod; Drug: ARV regimen
- Vesatolimod 10 or 12 mg (Cohort 6) (Experimental): Vesatolimod 10 or 12 mg for 127 days administered following overnight fasting, while continuing their existing ARV regimen. Participants will receive 3 administrations of 10 mg, followed by 7 administrations of 12 mg (after review of 10 mg safety data)
  Interventions: Drug: Vesatolimod; Drug: ARV regimen
- Vesatolimod 12 mg (Optional Cohort 7) (Experimental): Vesatolimod up to 12 mg for up to 127 days for up to 10 total doses administered following overnight fasting, while continuing their existing ARV regimen
  Interventions: Drug: Vesatolimod; Drug: ARV regimen
- Vesatolimod 6 mg with an acidic solution (Optional Cohort 8) (Experimental): Vesatolimod 6 mg for 127 days for up to 10 total doses administered with an acidic solution (cranberry juice), while continuing their existing ARV regimen
  Interventions: Drug: Vesatolimod; Drug: ARV regimen
- Vesatolimod up to 12 mg (Cohort 9) (Experimental): Vesatolimod up to 12 mg for 127 days for up to 10 total doses administered following a moderate-fat meal, after the review of the data from the highest tolerated fasted dose cohort while continuing their existing ARV regimen
  Interventions: Drug: Vesatolimod; Drug: ARV regimen
- Placebo (Cohorts 1-9) (Placebo Comparator): Placebo to match vesatolimod for 71 or 127 days, while continuing their existing ARV regimen
  Interventions: Drug: Placebo; Drug: ARV regimen

INTERVENTIONS:
Drug: Vesatolimod — Tablet(s) administered orally once every 2 weeks
  Other Names: GS-9620
  Arms: Vesatolimod 1 mg (Cohort 1); Vesatolimod 10 or 12 mg (Cohort 6); Vesatolimod 12 mg (Optional Cohort 7); Vesatolimod 2 mg (Cohort 2); Vesatolimod 4 mg (Cohort 3); Vesatolimod 6 mg (Cohort 4); Vesatolimod 6 mg with an acidic solution (Optional Cohort 8); Vesatolimod 8 mg (Cohort 5); Vesatolimod up to 12 mg (Cohort 9)
Drug: Placebo — Tablet(s) administered orally once every 2 weeks
  Arms: Placebo (Cohorts 1-9)
Drug: ARV regimen — Participants' current ARV regimen must be used in accordance with their prescribing information and may include the following: nucleoside/nucleotide reverse transcriptase inhibitors (NRTIs), raltegravir, dolutegravir, rilpivirine, and maraviroc.

SUMMARY:
The primary objectives of this study are to evaluate the safety and tolerability of escalating, multiple doses of vesatolimod (formerly GS-9620) in HIV-1 infected virologically suppressed adults on antiretroviral therapy (ART) and to evaluate the virologic effect of vesatolimod as measured by changes in plasma HIV-1 RNA.

ELIGIBILITY:
Key Inclusion Criteria:

* HIV-1 infection
* Aged ≥ 18 years at Pre-baseline/Day -13
* On antiretroviral (ARV) treatment for ≥ 12 consecutive months prior to Pre-Baseline/Day -13

  * The following agents are allowed as part of the current ARV regimen: NRTIs, raltegravir, dolutegravir, rilpivirine, and maraviroc
  * The following agents are NOT allowed as part of the current ARV regimen: HIV protease inhibitors (including low dose ritonavir), cobicistat-containing regimens, elvitegravir, efavirenz, etravirine, and nevirapine
  * A change in ARV regimen ≥ 45 days prior to baseline/Day 1 for reasons other than virologic failure (eg, tolerability, simplification, drug-drug interaction profile) is allowed
* Plasma HIV-1 RNA < 50 copies/mL at screening
* Documented plasma HIV-1 RNA levels < 50 copies/mL (according to the local assay being used) for ≥ 12 months preceding the screening visit (measured at least twice using a licensed assay with a lower limit of quantitation of at least 40 copies/mL)

  * Unconfirmed virologic elevations of ≥ 50 copies/mL (transient detectable viremia, or "blip") prior to screening are acceptable. (If the lower limit of detection of the local HIV-1 RNA assay is < 50 copies/mL, the plasma HIV-1 RNA level cannot exceed 50 copies/mL on two consecutive HIV-1 RNA tests)
  * If ART regimen is changed ≥ 60 days prior to Pre-Baseline/Day -13, plasma HIV-1 RNA <50 copies/mL at Pre-baseline/Day -13 visit is required
* No documented history of resistance to any components of the current ARV regimen
* Availability of a fully active alternative ARV regimen, in the opinion of the Investigator, in the event of discontinuation of the current ARV regimen with development of resistance
* Hgb ≥ 11.5 g/dL (males) or ≥ 11 g/dL (females)
* White blood cells (WBC) ≥ 4,000 cells/μL
* Platelets ≥ 150,000/mL
* Absolute neutrophil count (ANC) ≥ 1500 cells/μL
* CD4 count ≥ 400 cells/μL
* Albumin ≥ 3.9 g/dL
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2 × upper limit of the normal range (ULN)
* Estimated glomerular filtration rate ≥ 60 mL/min
* No autoimmune disease

Key Exclusion Criteria:

* Hepatitis B surface antigen (HBsAg) positive

  * Positive anti-HBs antibody and negative HBsAg results are acceptable
* Hepatitis C antibody (HCVAb) positive

  * Positive anti-HCV antibody and negative HCV polymerase chain reaction (PCR) results are acceptable
* Documented history of pre-ART CD4 nadir < 200 cells/µL

  * Unknown pre-ART CD4 nadir is acceptable
* A new AIDS-defining condition diagnosed within 90 days prior to screening
* Acute febrile illness within 35 days prior to pre-baseline/Day -13

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-01-29 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (8):
- United States (8):
  - Mills Clinical Research, Los Angeles, California
  - UCSD Antiviral Research Center (AVRC), San Diego, California
  - Midway Immunology & Research Center, Ft. Pierce, Florida
  - Orlando Immunology Center Recruiting, Orlando, Florida
  - Ohio State University Infectious Diseases Research, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Central Texas Clinical Research, Austin, Texas
  - Peter Shalit, MD, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Riddler S, Para M, Benson C, et al. Vesatolimod (GS-9620) is safe and pharmacodynamically active in HIV infected individuals [Oral presentation WEAA0304]. 10th International AIDS Society Conference on HIV Science (IAS 2019), 22-23 July 2019, Mexico City, Mexico
- [Derived] Riddler SA, Para M, Benson CA, Mills A, Ramgopal M, DeJesus E, Brinson C, Cyktor J, Jacobs J, Koontz D, Mellors JW, Laird GM, Wrin T, Patel H, Guo S, Wallin J, Boice J, Zhang L, Humeniuk R, Begley R, German P, Graham H, Geleziunas R, Brainard DM, SenGupta D. Vesatolimod, a Toll-like Receptor 7 Agonist, Induces Immune Activation in Virally Suppressed Adults Living With Human Immunodeficiency Virus-1. Clin Infect Dis. 2021 Jun 1;72(11):e815-e824. doi: 10.1093/cid/ciaa1534. PMID 33043969

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United States. The first participant was screened on 29 January 2015. The last study visit occurred on 14 February 2019.
Pre-assignment Details: 58 participants were screened.
Groups:
- Vesatolimod 1 mg (Cohort 1): Participants received vesatolimod 1 mg orally following 2-hour fast once every 2 weeks for 71 days for a total of 6 doses while continuing their existing antiretroviral (ARV) regimen in accordance with their prescribing information (the following agents were allowed: nucleoside/nucleotide reverse transcriptase inhibitors [NRTIs], raltegravir, dolutegravir, rilpivirine, and maraviroc).
- Vesatolimod 2 mg (Cohort 2): Participants received vesatolimod 2 mg orally following 2-hour fast once every 2 weeks for 71 days for a total of 6 doses while continuing their ARV regimen in accordance with their prescribing information (the following agents were allowed: NRTIs, raltegravir, dolutegravir, rilpivirine, and maraviroc).
- Vesatolimod 4 mg (Cohort 3): Participants received vesatolimod 4 mg orally following 2-hour fast once every 2 weeks for 71 days for a total of 6 doses while continuing their ARV regimen in accordance with their prescribing information (the following agents were allowed: NRTIs, raltegravir, dolutegravir, rilpivirine, and maraviroc).
- Vesatolimod 6 mg (Cohort 4): Participants received vesatolimod 6 mg orally following 2-hour fast once every 2 weeks for 127 days for a total of 10 doses, while continuing their ARV regimen in accordance with their prescribing information (the following agents were allowed: NRTIs, raltegravir, dolutegravir, rilpivirine, and maraviroc).
- Vesatolimod 8 mg (Cohort 5): Participants received vesatolimod 8 mg orally following overnight fasting once every 2 weeks for 127 days for a total of 10 doses, while continuing their ARV regimen in accordance with their prescribing information (the following agents were allowed: NRTIs, raltegravir, dolutegravir, rilpivirine, and maraviroc).
- Vesatolimod 10 or 12 mg (Cohort 6): Participants received vesatolimod 10 mg orally up to Day 43 for a total of 3 doses then vesatolimod 12 mg orally up to Day 127 for a total 7 doses following overnight fasting once every 2 weeks while continuing their existing ARV regimen in accordance with their prescribing information (the following agents were allowed: NRTIs, raltegravir, dolutegravir, rilpivirine, and maraviroc).
- Placebo: Participants received vesatolimod placebo orally once every 2 weeks for 71 days for a total of 6 doses or 127 days for a total of 10 doses while continuing their existing ARV regimen in accordance with their prescribing information (the following agents were allowed: NRTIs, raltegravir, dolutegravir, rilpivirine, and maraviroc).
Period: Overall Study
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Started | 6 | 6 | 6 | 6 | 6 | 6 | 12
Completed | 6 | 5 | 6 | 6 | 6 | 5 | 12
Not Completed | 0 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrew Consent | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug.
Groups:
- Vesatolimod 1 mg (Cohort 1): Participants received vesatolimod 1 mg orally following 2-hour fast once every 2 weeks for 71 days for a total of 6 doses while continuing their existing ARV regimen in accordance with their prescribing information (the following agents were allowed: NRTIs, raltegravir, dolutegravir, rilpivirine, and maraviroc).
- Vesatolimod 8 mg (Cohort 5): Participants received vesatolimod 8 mg orally following overnight fasting once every 2 weeks for 127 days for a total of 10 doses, while continuing their ARV regimen in accordance their prescribing information (the following agents were allowed: NRTIs, raltegravir, dolutegravir, rilpivirine, and maraviroc).
- Total: Total of all reporting groups
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (11.0) | 45 (10.7) | 52 (4.8) | 44 (9.3) | 45 (9.9) | 47 (17.5) | 45 (11.9) | 46 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 5
  Male | 6 | 5 | 6 | 6 | 3 | 5 | 12 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 5
  Not Hispanic or Latino | 5 | 4 | 6 | 6 | 4 | 6 | 12 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
  White | 6 | 6 | 6 | 5 | 5 | 6 | 12 | 46
HIV-1 RNA [Mean (Standard Deviation); unit: log10 copies/mL] | 1.28 (0.000) | 1.28 (0.000) | 1.30 (0.062) | 1.28 (0.000) | 1.28 (0.000) | 1.28 (0.000) | 1.28 (0.000) | 1.28 (0.022)
HIV-1 RNA Category [Count of Participants; unit: Participants]
  < 50 copies/ mL | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 48
  ≥ 50 copies/ mL | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Serious Adverse Events (SAEs) and Any Treatment-Emergent Adverse Events (AEs).
Time Frame: For Cohorts 1 to 3: First dose date up to 71 days plus 30 days; For Cohorts 4 to 6: First dose date up to 127 days plus 30 days; For placebo: First dose date up to 71 days plus 30 days or first dose date up to 127 days plus 30 days
Population: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
percentage of participants
  SAEs | 0.0 | 16.7 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  AEs | 66.7 | 66.7 | 33.3 | 66.7 | 83.3 | 66.7 | 75.0

2. Primary Outcome: Maximum Change From Baseline in Plasma Log10 HIV-1 RNA at Any Postdose Timepoint
Description: The maximum change from baseline in plasma Log10 HIV-1 RNA refers to the maximum change at any postdose timepoint up to Day 81 or Day 134 for placebo, Day 81 for Cohorts 1 to 3, and Day 134 for Cohorts 4 to 6.
Time Frame: For Cohorts 1 to 3: Baseline to Day 81; For Cohorts 4 to 6: Baseline to Day 134; For placebo: Baseline to Day 81 or Baseline to Day 134
Population: The Full Analysis Set included participants who were randomized and received at least 1 dose of study drug.
Measure: Mean (Standard Error); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
Log10 copies/mL | 0.06 (0.141) | 0.01 (0.018) | 0.10 (0.252) | 0.04 (0.092) | 0.00 (0.000) | 0.07 (0.073) | 0.42 (0.729)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 0.1498, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 0.0640, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 0.2807, Wilcoxon rank sum test
Statistical Analysis 4: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 0.1228, Wilcoxon rank sum test
Statistical Analysis 5: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 0.0289, Wilcoxon rank sum test
Statistical Analysis 6: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 0.5895, Wilcoxon rank sum test

3. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 2
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 2.
Time Frame: Baseline; Day 2
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 6 | 5
Log10 copies/mL |  |  |  | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
Statistical Analysis 1: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test

4. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 3
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 3.
Time Frame: Baseline; Day 3
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 12
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.091) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.01 (0.034)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 0.5557, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 0.5557, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 0.8288, Wilcoxon rank sum test
Statistical Analysis 4: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 0.5557, Wilcoxon rank sum test
Statistical Analysis 5: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 0.6056, Wilcoxon rank sum test
Statistical Analysis 6: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 0.5557, Wilcoxon rank sum test

5. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 5
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 5.
Time Frame: Baseline; Day 5
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 0 | 6
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | -0.03 (0.062) |  |  |  | 0.00 (0.000)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 0.4047, Wilcoxon rank sum test

6. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 8
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 8.
Time Frame: Baseline; Day 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 12
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | -0.03 (0.068) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 0.1556, Wilcoxon rank sum test
Statistical Analysis 4: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 5: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 6: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test

7. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 11
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 11.
Time Frame: Baseline; Day 11
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 6 | 5 | 0 | 0 | 0 | 6
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | -0.03 (0.068) |  |  |  | 0.00 (0.000)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 0.3613, Wilcoxon rank sum test

8. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 15
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 15.
Time Frame: Baseline; Day 15
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 12
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | -0.03 (0.062) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 0.1949, Wilcoxon rank sum test
Statistical Analysis 4: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 5: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 6: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test

9. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 17
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 17.
Time Frame: Baseline; Day 17
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 0 | 6
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | 0.01 (0.117) |  |  |  | 0.00 (0.000)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test

10. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 19
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 19.
Time Frame: Baseline; Day 19
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Groups:
- Vesatolimod 1 mg (Cohort 1): Participants received vesatolimod 1 mg tablet orally following 2-hour fast once every 2 weeks for 71 days for a total of 6 doses while continuing their existing ARV regimen in accordance with their prescribing information (the following agents were allowed: NRTIs, raltegravir, dolutegravir, rilpivirine, and maraviroc).
- Vesatolimod 2 mg (Cohort 2): Participants received vesatolimod 2 mg tablet orally following 2-hour fast once every 2 weeks for 71 days for a total of 6 doses while continuing their ARV regimen in accordance with their prescribing information (the following agents were allowed: NRTIs, raltegravir, dolutegravir, rilpivirine, and maraviroc).
- Vesatolimod 4 mg (Cohort 3): Participants received vesatolimod 4 mg tablet orally following 2-hour fast once every 2 weeks for 71 days for a total of 6 doses while continuing their ARV regimen in accordance with their prescribing information (the following agents were allowed: NRTIs, raltegravir, dolutegravir, rilpivirine, and maraviroc).
- Vesatolimod 6 mg (Cohort 4): Participants received vesatolimod 6 mg tablet orally following 2-hour fast once every 2 weeks for 127 days for a total of 10 doses while continuing their ARV regimen in accordance with their prescribing information (the following agents were allowed: NRTIs, raltegravir, dolutegravir, rilpivirine, and maraviroc).
- Vesatolimod 8 mg (Cohort 5): Participants received vesatolimod 8 mg tablet following overnight fasting once every 2 weeks for 127 days for a total of 10 doses while continuing their ARV regimen in accordance with their prescribing information (the following agents were allowed: NRTIs, raltegravir, dolutegravir, rilpivirine, and maraviroc).
- Vesatolimod 10 or 12 mg (Cohort 6): Participants received vesatolimod 10 mg up to Day 43 for a total of 3 doses then vesatolimod 12 mg up to 12 mg for a total 7 doses following overnight fasting once every 2 weeks while continuing their existing ARV regimen in accordance with their prescribing information (the following agents were allowed: NRTIs, raltegravir, dolutegravir, rilpivirine, and maraviroc).
- Placebo: Participants received vesatolimod placebo once every 2 weeks for 71 days for a total of 6 doses or 127 days for a total of 10 doses while continuing their existing ARV regimen in accordance with their prescribing information (the following agents were allowed: NRTIs, raltegravir, dolutegravir, rilpivirine, and maraviroc).
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 0 | 6
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | -0.03 (0.062) |  |  |  | 0.00 (0.000)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 0.4047, Wilcoxon rank sum test

11. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 22
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 22.
Time Frame: Baseline; Day 22
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 12
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | 0.02 (0.037) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 0.1556, Wilcoxon rank sum test
Statistical Analysis 4: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 5: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 6: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test

12. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 25
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 25.
Time Frame: Baseline; Day 25
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 0 | 0 | 0 | 6
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | -0.03 (0.062) |  |  |  | 0.00 (0.000)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 0.4047, Wilcoxon rank sum test

13. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 29
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 29.
Time Frame: Baseline; Day 29
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 12
Log10 copies/mL | 0.01 (0.018) | 0.00 (0.000) | 0.02 (0.112) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 0.1949, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 0.4278, Wilcoxon rank sum test
Statistical Analysis 4: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 5: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 6: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test

14. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 31
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 31.
Time Frame: Baseline; Day 31
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 5 | 6 | 0 | 6 | 6 | 10
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | -0.03 (0.062) |  | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.014)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 0.5186, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 0.5716, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 0.1869, Wilcoxon rank sum test
Statistical Analysis 4: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 0.5186, Wilcoxon rank sum test
Statistical Analysis 5: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 0.5186, Wilcoxon rank sum test

15. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 33
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 33.
Time Frame: Baseline; Day 33
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 5 | 6 | 0 | 0 | 0 | 5
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | -0.03 (0.062) |  |  |  | 0.01 (0.028)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 0.3613, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 0.4237, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 0.2230, Wilcoxon rank sum test

16. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 36
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 36
Time Frame: Baseline; Day 36
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 12
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | -0.03 (0.062) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.16 (0.500)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 0.3456, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 0.3971, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 0.1301, Wilcoxon rank sum test
Statistical Analysis 4: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 0.3456, Wilcoxon rank sum test
Statistical Analysis 5: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 0.3456, Wilcoxon rank sum test
Statistical Analysis 6: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 0.3456, Wilcoxon rank sum test

17. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 39
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 39
Time Frame: Baseline; Day 39
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 5 | 6 | 0 | 0 | 0 | 6
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | 0.04 (0.190) |  |  |  | 0.25 (0.620)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 0.4047, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 0.4652, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 0.5993, Wilcoxon rank sum test

18. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 43
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 43
Time Frame: Baseline; Day 43
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 12
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | -0.03 (0.062) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 0.1949, Wilcoxon rank sum test
Statistical Analysis 4: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 5: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 6: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test

19. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 45
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit pn Day 45
Time Frame: Baseline; Day 45
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 5 | 6 | 0 | 6 | 6 | 9
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | -0.03 (0.062) |  | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 0.2763, Wilcoxon rank sum test
Statistical Analysis 4: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 5: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test

20. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 47
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 47
Time Frame: Baseline; Day 47
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 5 | 5 | 0 | 0 | 0 | 6
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | 0.07 (0.249) |  |  |  | 0.00 (0.000)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test

21. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 50
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 50.
Time Frame: Baseline; Day 50
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 12
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | -0.03 (0.062) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 0.1949, Wilcoxon rank sum test
Statistical Analysis 4: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 5: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 6: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test

22. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 53
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 53
Time Frame: Baseline; Day 53
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 5 | 6 | 0 | 0 | 0 | 6
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | 0.01 (0.126) |  |  |  | 0.00 (0.000)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test

23. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 57
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 57.
Time Frame: Baseline; Day 57
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 11
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | 0.03 (0.165) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.03 (0.097)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 0.5383, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 0.5896, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 0.8207, Wilcoxon rank sum test
Statistical Analysis 4: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 0.5383, Wilcoxon rank sum test
Statistical Analysis 5: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 0.5383, Wilcoxon rank sum test
Statistical Analysis 6: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 0.5383, Wilcoxon rank sum test

24. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 58
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 58.
Time Frame: Baseline; Day 58
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 6 | 5
Log10 copies/mL |  |  |  | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
Statistical Analysis 1: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test

25. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 59
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 59.
Time Frame: Baseline; Day 59
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 11
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | -0.01 (0.081) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.07 (0.190)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 0.3237, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 0.3755, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 0.4577, Wilcoxon rank sum test
Statistical Analysis 4: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 0.3237, Wilcoxon rank sum test
Statistical Analysis 5: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 0.3237, Wilcoxon rank sum test
Statistical Analysis 6: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 0.3237, Wilcoxon rank sum test

26. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 61
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 61.
Time Frame: Baseline; Day 61
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 5 | 6 | 0 | 0 | 0 | 6
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | 0.01 (0.126) |  |  |  | 0.03 (0.081)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 0.4047, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 0.4652, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 0.7526, Wilcoxon rank sum test

27. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 64
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 64.
Time Frame: Baseline; Day 64
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 5 | 5 | 6 | 6 | 6 | 6 | 11
Log10 copies/mL | 0.07 (0.154) | 0.01 (0.019) | 0.07 (0.249) | 0.00 (0.000) | 0.00 (0.000) | 0.02 (0.041) | 0.02 (0.072)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 0.5546, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 0.6937, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 0.8207, Wilcoxon rank sum test
Statistical Analysis 4: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 0.5383, Wilcoxon rank sum test
Statistical Analysis 5: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 0.5383, Wilcoxon rank sum test
Statistical Analysis 6: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 0.7878, Wilcoxon rank sum test

28. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 67
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 67.
Time Frame: Baseline; Day 67
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 5 | 6 | 0 | 0 | 0 | 6
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | 0.04 (0.194) |  |  |  | 0.00 (0.000)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test

29. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 71
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 71.
Time Frame: Baseline; Day 71
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 12
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | 0.02 (0.140) | 0.00 (0.000) | 0.00 (0.000) | 0.02 (0.056) | 0.00 (0.000)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 4: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 5: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 0.1949, Wilcoxon rank sum test

30. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 73
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 73.
Time Frame: Baseline; Day 73
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 5 | 6 | 0 | 6 | 6 | 10
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | 0.01 (0.112) |  | 0.00 (0.000) | 0.00 (0.000) | 0.04 (0.136)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 0.5186, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 0.5716, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 0.6908, Wilcoxon rank sum test
Statistical Analysis 4: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 0.5186, Wilcoxon rank sum test
Statistical Analysis 5: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 0.5186, Wilcoxon rank sum test

31. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 75
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 75.
Time Frame: Baseline; Day 75
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 5 | 6 | 0 | 0 | 0 | 6
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | -0.03 (0.062) |  |  |  | 0.00 (0.000)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 0.4047, Wilcoxon rank sum test

32. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 78
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 78.
Time Frame: Baseline; Day 78
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 11
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | -0.03 (0.062) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.19 (0.635)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 0.5383, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 0.5896, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 0.1784, Wilcoxon rank sum test
Statistical Analysis 4: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 0.5383, Wilcoxon rank sum test
Statistical Analysis 5: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 0.5383, Wilcoxon rank sum test
Statistical Analysis 6: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 0.5383, Wilcoxon rank sum test

33. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 81
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 81.
Time Frame: Baseline; Day 81
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 5 | 5 | 0 | 0 | 0 | 6
Log10 copies/mL | 0.00 (0.000) | 0.00 (0.000) | -0.03 (0.071) |  |  |  | 0.00 (0.000)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test

34. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 85
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 85.
Time Frame: Baseline; Day 85
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Groups:
- Vesatolimod 2 mg (Cohort 2): Participants received vesatolimod 2 mg orally following 2-hour fast once every 2 weeks for 71 days for a total of 6 doses while continuing their ARV regimen in accordance with their prescribing (the following agents were allowed: NRTIs, raltegravir, dolutegravir, rilpivirine, and maraviroc).
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 6 | 6
Log10 copies/mL |  |  |  | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.03 (0.075)
Statistical Analysis 1: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 0.4047, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 0.4047, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 0.4047, Wilcoxon rank sum test

35. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 87
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 87.
Time Frame: Baseline; Day 87
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 6 | 4
Log10 copies/mL |  |  |  |  | 0.00 (0.000) | 0.00 (0.000) | 0.19 (0.385)
Statistical Analysis 1: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 0.3074, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 0.3074, Wilcoxon rank sum test

36. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 92
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 92.
Time Frame: Baseline; Day 92
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 6 | 6
Log10 copies/mL |  |  |  | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.11 (0.261)
Statistical Analysis 1: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 0.4047, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 0.4047, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 0.4047, Wilcoxon rank sum test

37. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 99
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 99.
Time Frame: Baseline; Day 99
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 6 | 6
Log10 copies/mL |  |  |  | 0.00 (0.000) | 0.00 (0.000) | 0.03 (0.062) | 0.07 (0.142)
Statistical Analysis 1: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 0.1757, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 0.1757, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 0.5993, Wilcoxon rank sum test

38. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 101
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 101.
Time Frame: Baseline; Day 101
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 5 | 6 | 0 | 6 | 6 | 10
Log10 copies/mL | 0.02 (0.049) | 0.00 (0.000) | 0.00 (0.102) |  | 0.00 (0.000) | 0.00 (0.000) | 0.05 (0.173)
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 0.8504, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 0.5716, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 0.6908, Wilcoxon rank sum test
Statistical Analysis 4: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 0.5186, Wilcoxon rank sum test
Statistical Analysis 5: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 0.5186, Wilcoxon rank sum test

39. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 106
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 106.
Time Frame: Baseline; Day 106
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 6 | 6
Log10 copies/mL |  |  |  | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.10 (0.250)
Statistical Analysis 1: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 0.4047, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 0.4047, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 0.4047, Wilcoxon rank sum test

40. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 113
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 113.
Time Frame: Baseline; Day 113
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 6 | 6
Log10 copies/mL |  |  |  | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.09 (0.218)
Statistical Analysis 1: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 0.4047, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 0.4047, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 0.4047, Wilcoxon rank sum test

41. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 115
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 115.
Time Frame: Baseline; Day 115
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 6 | 4
Log10 copies/mL |  |  |  |  | 0.00 (0.000) | 0.00 (0.000) | 0.08 (0.156)
Statistical Analysis 1: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 0.3074, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 0.3074, Wilcoxon rank sum test

42. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 120
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 120.
Time Frame: Baseline; Day 120
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 6 | 6
Log10 copies/mL |  |  |  | 0.04 (0.092) | 0.00 (0.000) | 0.00 (0.000) | 0.01 (0.018)
Statistical Analysis 1: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 0.4047, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 0.4047, Wilcoxon rank sum test

43. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 127
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 127.
Time Frame: Baseline; Day 127
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 5 | 6
Log10 copies/mL |  |  |  | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
Statistical Analysis 1: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 1.0000, Wilcoxon rank sum test

44. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 128
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 128.
Time Frame: Baseline; Day 128
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 5 | 6
Log10 copies/mL |  |  |  | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.06 (0.129)
Statistical Analysis 1: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 0.1757, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 0.1757, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 0.2230, Wilcoxon rank sum test

45. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 129
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 129.
Time Frame: Baseline; Day 129
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 5 | 6
Log10 copies/mL |  |  |  | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.03 (0.062)
Statistical Analysis 1: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 0.4047, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 0.4047, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 0.4652, Wilcoxon rank sum test

46. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 134
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 134.
Time Frame: Baseline; Day 134
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 5 | 6
Log10 copies/mL |  |  |  | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.09 (0.215)
Statistical Analysis 1: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 0.4047, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 0.4047, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 0.4652, Wilcoxon rank sum test

47. Secondary Outcome: Change From Baseline in Plasma Log10 HIV-1 RNA at Day 157
Description: Change from baseline in plasma log10 HIV-1 RNA refers to change from baseline at a postbaseline visit on Day 157.
Time Frame: Baseline; Day 157
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 5 | 6
Log10 copies/mL |  |  |  | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.13 (0.254)
Statistical Analysis 1: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 0.1757, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 0.1757, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 0.2230, Wilcoxon rank sum test

48. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA ≥ 50 Copies/mL at Postdose 1 on Day 1
Time Frame: Postdose 1 on Day 1
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

49. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA ≥ 50 Copies/mL at PostDose 2 on Day 15
Time Frame: PostDose 2 on Day 15
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 12
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

50. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA ≥ 50 Copies/mL at PostDose 3 on Day 29
Time Frame: PostDose 3 on Day 29
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 12
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 8.3
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 4: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 5: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 6: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact

51. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA ≥ 50 Copies/mL at PostDose 4 on Day 43
Time Frame: PostDose 4 on Day 43
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 12
percentage of participants | 0.0 | 0.0 | 16.7 | 0.0 | 0.0 | 0.0 | 0.0
Statistical Analysis 1: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 0.3333, Fisher Exact

52. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA ≥ 50 Copies/mL at PostDose 5 on Day 57
Time Frame: PostDose 5 on Day 57
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 11
percentage of participants | 0.0 | 0.0 | 16.7 | 0.0 | 0.0 | 0.0 | 9.1
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 4: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 5: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 6: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact

53. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA ≥ 50 Copies/mL at PostDose 6 on Day 71
Time Frame: PostDose 6 on Day 71
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 6 | 5 | 6 | 5 | 6 | 6 | 11
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 9.1
Statistical Analysis 1: Comparison: Vesatolimod 1 mg (Cohort 1) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Vesatolimod 2 mg (Cohort 2) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 3: Comparison: Vesatolimod 4 mg (Cohort 3) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 4: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 5: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 6: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact

54. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA ≥ 50 Copies/mL at PostDose 7 on Day 85
Time Frame: PostDose 7 on Day 85
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 6 | 6
percentage of participants |  |  |  | 0.0 | 0.0 | 0.0 | 16.7
Statistical Analysis 1: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 3: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact

55. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA ≥ 50 Copies/mL at PostDose 8 on Day 99
Time Frame: PostDose 8 on Day 99
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 6 | 6 | 6
percentage of participants |  |  |  | 0.0 | 0.0 | 0.0 | 16.7
Statistical Analysis 1: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 3: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact

56. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA ≥ 50 Copies/mL at PostDose 9 on Day 113
Time Frame: PostDose 9 on Day 113
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 6 | 6 | 6
percentage of participants |  |  |  | 0.0 | 0.0 | 0.0 | 0.0

57. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA ≥ 50 Copies/mL at PostDose 10 on Day 127
Time Frame: PostDose 10 on Day 127
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 5 | 6
percentage of participants |  |  |  | 0.0 | 0.0 | 0.0 | 16.7
Statistical Analysis 1: Comparison: Vesatolimod 6 mg (Cohort 4) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Vesatolimod 8 mg (Cohort 5) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 3: Comparison: Vesatolimod 10 or 12 mg (Cohort 6) vs Placebo; Test type: Other; p = 1.0000, Fisher Exact

ADVERSE EVENTS:
Time Frame: For Cohorts 1 to 3: First dose date up to 71 days plus 30 days; For Cohorts 4 to 6: First dose date up to 127 days plus 30 days; For placebo: First dose date up to 71 days plus 30 days or first dose date up to 127 days plus 30 days
Description: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug.
Arm/Group | Vesatolimod 1 mg (Cohort 1) | Vesatolimod 2 mg (Cohort 2) | Vesatolimod 4 mg (Cohort 3) | Vesatolimod 6 mg (Cohort 4) | Vesatolimod 8 mg (Cohort 5) | Vesatolimod 10 or 12 mg (Cohort 6) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 4/6 | 4/6 | 2/6 | 4/6 | 5/6 | 4/6 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vesatolimod 1 mg (Cohort 1) (N=6) | Vesatolimod 2 mg (Cohort 2) (N=6) | Vesatolimod 4 mg (Cohort 3) (N=6) | Vesatolimod 6 mg (Cohort 4) (N=6) | Vesatolimod 8 mg (Cohort 5) (N=6) | Vesatolimod 10 or 12 mg (Cohort 6) (N=6) | Placebo (N=12)
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vesatolimod 1 mg (Cohort 1) (N=6) | Vesatolimod 2 mg (Cohort 2) (N=6) | Vesatolimod 4 mg (Cohort 3) (N=6) | Vesatolimod 6 mg (Cohort 4) (N=6) | Vesatolimod 8 mg (Cohort 5) (N=6) | Vesatolimod 10 or 12 mg (Cohort 6) (N=6) | Placebo (N=12)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erythema of eyelid (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Scleral hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 1 | 1 | 1
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Early satiety (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 1 | 1 | 0 | 3 | 3
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Sluggishness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bone abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Proctitis gonococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Syphilis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinea cruris (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Exposure to communicable disease (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eyelid contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 2
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Slow speech (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Genital lesion (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 1
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pseudofolliculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2019-01-16): https://cdn.clinicaltrials.gov/large-docs/01/NCT02858401/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT02858401/SAP_001.pdf